CLINICAL TRIAL: NCT01114451
Title: A Randomized Controlled Trial of Early Versus Delayed Skin Staple Removal Following Cesarean Delivery in the Obese Patient
Brief Title: Early Versus Delayed Skin Staple Removal Following Cesarean Delivery in the Obese Patient
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding limits exceeded prior to complete enrollment.
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002576
Record Dates: First submitted 2010-04-16; First posted 2010-05-03 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Wound Complications; Obesity
Keywords: Cesarean delivery; Obesity; Skin staples; Wound complications
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Staple Removal (Experimental): Skin staple removal on post-operative day #3
  Interventions: Procedure: Removal of surgical skin staples
- Delayed Staple Removal (Experimental): Skin staple removal on post-operative day 7-10
  Interventions: Procedure: Removal of surgical skin staples

INTERVENTIONS:
Procedure: Removal of surgical skin staples — Skin staples will be removed using standard technique with subsequent placement of steri-trips

SUMMARY:
Whenever a person has a cesarean section there is a risk that there will be a problem with healing of the wound. The most common type of wound healing problem is separation and opening of the skin and fatty tissue just beneath the skin. This type of wound healing problem happens more often when the patient has a high body weight. In most cases, metal staples are used to bring the skin together to close the wound. Usually, the staples are left in place for a longer time when the woman is heavy, in hopes of decreasing the chance of wound healing problems. But it is not known if leaving the staples in for a longer time is actually helpful. In some cases, leaving the staples in longer may cause more pain and will require you to see the doctor again to get the staples taken out. The purpose of this study is to see if there is any difference in how the wound heals in heavy women after cesarean section when the skin staples are removed after a short period of time versus a long period of time.

DETAILED DESCRIPTION:
Cesarean delivery in the obese gravida is associated with numerous perioperative risks, the most frequent of which is postoperative wound disruption, with a mean incidence of 15%. With the exception of closure of the subcutaneous adipose layer, other useful measures to decrease wound complications in the obese gravida have either not been studied or lack sufficient evidence upon which to base a recommendation.

One such intervention is the delayed removal of surgical skin staples. Skin staplers, which were first introduced in the 1980's, were "grandfathered" through the United States Food and Drug Administration (FDA) approval process, and have since become a widely utilized technique for skin closure. Although neither the FDA nor device manufacturers make a specific recommendation, skin staples are commonly left in situ anywhere from 3 - 10 days.

The physiologic rationale for delayed staple removal is unclear. Wound healing involves four main stages including hemostasis, inflammation, granulation, and remodeling. Each phase can be further broken down into overlapping steps. Reapproximation of the skin edges with staples enables epithelialization, resulting in wound closure by a thin layer of cells by 48 hours post-operatively. Although overall wound healing appears to be delayed in the setting of obesity, whether the specific process of epithelialization is affected is unknown. Therefore, there may not be a physiologic basis for delaying staple removal in obese women.

Furthermore, delayed staple removal has potentially negative effects on patient care that may not be balanced by clinical benefits. Delayed staple removal may be associated with prolongation of patient discomfort, additional clinical visits and increased associated costs. These issues caused us to question whether the practice of delayed skin staple removal in obese women is warranted.

Therefore, this clinical trial is designed to compare wound healing outcomes after cesarean following early (postoperative day #3) versus delayed (postoperative day #7 - 10) skin staple removal in the obese patient.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery
* Body Mass Index ≥ 30 kg/m2
* Transverse (Pfannenstiel or Joel-Cohen) skin incision
* Subcutaneous wound depth ≥ 2 cm
* Surgical staple skin closure

Exclusion Criteria:

* Vertical skin incision
* Non-staple skin closure
* Wound complication (superficial dehiscence, abscess, seroma, hematoma, cellulitis)
* Any complication necessitating prolonged hospitalization

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with a superficial wound disruption as a measure of efficacy. | 7-10 days after surgery
  Any separation of the wound edge measuring greater than 1 cm that occurs from the time of staple placement to final wound assessment which occurs at 7-10 days after surgery.

SECONDARY OUTCOMES:
Number of participants who develop a wound seroma. | 6 weeks after surgery
  A collection of fluid within the subcutaneous fatty tissue layer.
Number of participants who develop a hematoma of the wound. | 6 weeks after surgery
  A collection of clotted blood within the subcutaneous tissues.
Number of participants who develop a surgical site infection | 6 weeks after surgery
  Infection involving only skin or subcutaneous tissue of the incision which occurs within 30 days after the operation.
Frequency of Visual Analogue Pain Score | 7-10 days after surgery
  Patient rating of pain on a 1-10 scale as assessed at the 7-10 day postoperative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Francis S Nuthalapaty, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States

REFERENCES:
- [Background] Nuthalapaty FS, Rouse DJ. The impact of obesity on obstetrical practice and outcome. Clin Obstet Gynecol. 2004 Dec;47(4):898-913; discussion 980-1. doi: 10.1097/01.grf.0000135358.34673.48. No abstract available. PMID 15596944
- [Background] Sarsam SE, Elliott JP, Lam GK. Management of wound complications from cesarean delivery. Obstet Gynecol Surv. 2005 Jul;60(7):462-73. doi: 10.1097/01.ogx.0000166603.43959.aa. PMID 15995563
- [Background] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Background] American College of Obstetricians and Gynecologists. ACOG Committee Opinion number 315, September 2005. Obesity in pregnancy. Obstet Gynecol. 2005 Sep;106(3):671-5. doi: 10.1097/00006250-200509000-00054. PMID 16135613
- [Background] Walsh C, Scaife C, Hopf H. Prevention and management of surgical site infections in morbidly obese women. Obstet Gynecol. 2009 Feb;113(2 Pt 1):411-5. doi: 10.1097/AOG.0b013e3181945625. No abstract available. PMID 19155915